CLINICAL TRIAL: NCT03033134
Title: A Study to Evaluate the Safety and Effectiveness of the Left Atrial Appendage Closure Therapy Using BSJ003W for Patients With Non-valvular Atrial Fibrillation at Increased Risk of ThromboEmbolism in Japanese Medical Environment (SALUTE)
Brief Title: A Study to Evaluate the Safety and Effectiveness of the Left Atrial Appendage Closure Therapy Using BSJ003W
Acronym: SALUTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Japan K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S6001
Record Dates: First submitted 2017-01-16; First posted 2017-01-26 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation Non-Rheumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- BSJ003W (Experimental): BSJ003W implant group
  Interventions: Device: BSJ003W

INTERVENTIONS:
Device: BSJ003W — BSJ003W implant

SUMMARY:
The purpose of this study is to confirm the safety and effectiveness of the BSJ003W in Japanese patients with non-valvular atrial fibrillation at increased risk of thromboembolism in Japanese Clinical environment

ELIGIBILITY:
Inclusion Criteria:

1. The subject is Japanese, over 20 years old and provides written informed consent to participate in the trial
2. The subject has documented paroxysmal, persistent or permanent non-valvular atrial fibrillation
3. The subject has a calculated CHA2DS2-VASc score of 2 or greater and is recommended for long-term oral anti-coagulation therapy
4. The subject is deemed by their physicians to be suitable for anticoagulant therapy and have an appropriate rationale to seek a non-pharmacologic alternative to warfarin
5. The subject is eligible to come off warfarin therapy if the LAA (left atrial appendage) is sealed (i.e. the subject has no other conditions that would require warfarin therapy).

Exclusion Criteria:

1. The subject has a prior stroke (ischemic or hemorrhagic) or transient ischemic attack within the 90 days prior to consent
2. The subject has had a myocardial infarction either non-ST elevation or ST elevation myocardial infarction within 90 days prior to consent with or without intervention
3. The subject had or is planning to have any cardiac (e.g. cardioversion, coronary angiogram, percutaneous coronary intervention, cardiac ablation, etc.) or non-cardiac invasive or surgical procedure (e.g. cataract surgery, endoscopy, etc.) within 30 days prior or 45 days after the BSJ003W implant
4. The subject has a history of atrial septal repair or has an atrial septal defect/persistent foramen ovale device
5. The subject has an implanted mechanical valve prosthesis in any position
6. The subject currently New York Heart Association class IV congestive heart failure
7. The subject is contraindicated to aspirin
8. The subject is contraindicated or seriously allergic to thienopyridine
9. The subject is of childbearing potential and is, or plans to become pregnant during the time of the study
10. The subject is not able and willing to return for required follow-up visits and examinations
11. Subjects who are currently enrolled in another investigational study (of which primary endpoint follow-up have not been completed yet).
12. The subject has other reason not to be eligible for this study per investigators' discretion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazutaka Aonuma, Principal Investigator — Tsukuba University Hospital; Shigeru Saito, Principal Investigator — Shonankamakura General Hospital
Locations (10):
- Japan (10):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Iwate Medical University Hospital, Morioka, Iwate
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Tokyo Medical and Dental University Medical Hospital, Bunkyo-ku, Tokyo
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No
The confidentiality of records/data obtained in the trial will remain anonymous for analysis and publication.
  The information and data, obtained from the trial is used without personal identification

REFERENCES:
- [Derived] Aonuma K, Yamasaki H, Nakamura M, Matsumoto T, Takayama M, Ando K, Hirao K, Goya M, Morino Y, Hayashida K, Kusano K, Gomi Y, Main ML, Uchida T, Saito S. Efficacy and Safety of Left Atrial Appendage Closure With WATCHMAN in Japanese Nonvalvular Atrial Fibrillation Patients - Final 2-Year Follow-up Outcome Data From the SALUTE Trial. Circ J. 2020 Jul 22;84(8):1237-1243. doi: 10.1253/circj.CJ-20-0196. Epub 2020 Jun 26. PMID 32595176

RESULTS

PARTICIPANT FLOW:
Groups:
- Implant (ITT): BSJ003W implant group (ITT) : 42 subjects
- Roll-in: 12 Roll-in subjects
Period: Overall Study
Arm/Group | Implant (ITT) | Roll-in
Started | 42 | 12
6-month Primary Endpoints | 42 | 12
Completed | 0 | 0
Not Completed | 42 | 12

BASELINE CHARACTERISTICS:
Groups:
- Implant (ITT): Implant (ITT) group: 42 subjects
- Roll-in: Roll-in group: 12 subjects
- Total: Total of all reporting groups
Arm/Group | Implant (ITT) | Roll-in | Total
Number analyzed (Participants) | 42 | 12 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (8.8) | 70.6 (7.4) | 72.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 35 | 10 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 42 | 12 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 42 | 12 | 54
CHA2DS2-VASc score [Mean (Standard Deviation); unit: units on a scale] — CHA2DS2-VASc score is recommended to assess stroke risk. CHA2DS2-VASc score is calculated by the summed of the following factors; C:1: Congestive Heart Failure/ LV dysfunction, H:1: Hypertension, A:2: Age >75, D:1: Diabetes, S:2: Stroke/ TIA, V:1: Vascular disease, A:1: Age 65-74, Sc:1: Female.
  Total Score range: 0-9. Higher score indicates the higher stroke risk.
  units on a scale | 3.6 (1.6) | 3.5 (1.6) | 3.6 (1.6)
Atrial Fibrillation pattern [Count of Participants; unit: Participants]
  Documented Paroxysmal | 15 | 5 | 20
  Documented Persistent | 9 | 3 | 12
  Documented Permanent | 18 | 4 | 22
HAS-BLED score [Mean (Standard Deviation); unit: units on a scale] — HAS-BLED score is a Bleeding risk scores to quantify hemorrhage risk. HAS-BLED score is calculated by the summed of the following factors; H: Hypertension, A: Abnormal renal function, Abnormal liver function, S: Stroke, B: Bleeding, L: Labile INRs, E: Elderly > 65 years, D: Drugs (NSAIDs) or Alcohol.
  Total Score Range: 0-9. Higher score indicates higher bleeding risk.
  units on a scale | 2.9 (1.1) | 3.1 (1.1) | 3.0 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complications; One of the Following Events
Description: All-cause death, ischemic stroke, systemic embolism, or device- or procedure- related events requiring open cardiac surgery or major endovascular intervention such as pseudoaneurysm repair, arteriolar-venular fistula repair, or other major endovascular repair.
Time Frame: Between the time of implant and within 7 days following the procedure or by hospital discharge, whichever is later
Measure: Count of Participants; unit: Participants
Groups:
- Roll-in: Roll-in cohort
Arm/Group | Implant (ITT) | Roll-in
Number analyzed (Participants) | 42 | 12
Participants | 0 | 0

2. Primary Outcome: Number of Participants With One of the Following Events: Stroke (All/ Ischemic/ Hemorrhagic), Systemic Embolism and Cardiovascular(CV) Death (Including Unexplained Cause)
Description: The occurrence of composite events including stroke (all/ ischemic/ hemorrhagic), systemic embolism and cardiovascular death (including unexplained cause) till 6-month post implant
Time Frame: 24-month
Population: Data collected from Roll-in subjects was analyzed separately from those data collected from ITT cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Roll-in: Roll-in cohort: 12 subjects
Arm/Group | Implant (ITT) | Roll-in
Number analyzed (Participants) | 42 | 12
Participants
  Ischemic stroke | 3 | 1
  Hemorrhagic stroke | 0 | 0
  Systemic embolism | 0 | 0
  Cardiovascular death | 1 | 0

3. Primary Outcome: The Rate of Effective Left Atrial Appendage (LAA) Closure
Description: The effective LAA closure is defined as peri-device flow <= 5mm demonstrated by TEE.
  TEE measurements will be assessed by an independent Core Laboratory.
Time Frame: 45-day, 6-month, 12-month
Population: Data collected from Roll-in subjects was analyzed separately from those data collected from ITT cohort.
  One subject in Roll-in cohort at 6-month was not able to assessed by the Core laboratory due to the quality of the images
Measure: Count of Participants; unit: Participants
Arm/Group | Implant (ITT) | Roll-in
Number analyzed (Participants) | 42 | 12
Participants
  At 45-day | 42 | 12
  At 6-month | 42 | 11
  At 12-month: number analyzed (Participants) | 41 | 11
  At 12-month | 41 | 11

4. Secondary Outcome: Number of Participants With Major Bleeding
Description: Major bleeding is defined as per BARC bleeding definition type 3 or 5.
  Type 3 Type 3a: Overt bleeding plus hemoglobin drop of 3 to 5 g/dL* (provided hemoglobin drop is related to bleed), Any transfusion with overt bleeding
  Type 3b: Overt bleeding plus hemoglobin drop 5 g/dL* (provided hemoglobin drop is related to bleed) Cardiac tamponade, Bleeding requiring surgical intervention for control (excluding dental/nasal/skin/hemorrhoid), Bleeding requiring intravenous vasoactive agents
  Type 3c: Intracranial hemorrhage (does not include microbleeds or hemorrhagic transformation, does include intraspinal), Subcategories confirmed by autopsy or imaging or lumbar puncture Intraocular bleed compromising vision
  Type 5: fatal bleeding Type 5a: Probable fatal bleeding; no autopsy or imaging confirmation but clinically suspicious Type 5b: Definite fatal bleeding; overt bleeding or autopsy or imaging confirmation
Time Frame: 24-month
Population: Data collected from Roll-in subjects was analyzed separately from those data collected from ITT cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Implant (ITT) | Roll-in
Number analyzed (Participants) | 42 | 12
Participants | 2 | 2

5. Secondary Outcome: Number of Participants With Clinically Overt Non-fatal Bleeding
Description: Clinically overt non-fatal bleeding is defined as per BARC bleeding definition type 2.
  Type 2: any overt, actionable sign of hemorrhage (eg, more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for type 3, 4, or 5 but does meet at least one of the following criteria: (1) requiring nonsurgical, medical intervention by a healthcare professional, (2) leading to hospitalization or increased level of care, or (3) prompting evaluation
Time Frame: 24-month
Measure: Count of Participants; unit: Participants
Arm/Group | Implant (ITT) | Roll-in
Number analyzed (Participants) | 42 | 12
Participants | 3 | 0

6. Secondary Outcome: Number of Participants With Ischemic Stroke or Systemic Embolism
Description: The occurrence of ischemic stroke or systemic embolism (excluding 7 days after implanting or day after hospital discharge whichever is the later)
Time Frame: 24-month
Population: Data collected from Roll-in subjects was analyzed separately from those data collected from ITT cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Implant (ITT): Implant (ITT): 42 subjects
Arm/Group | Implant (ITT) | Roll-in
Number analyzed (Participants) | 42 | 12
Participants
  Ischemic stroke | 3 | 1
  Systemic embolism | 0 | 0

7. Other Pre Specified Outcome: Technical Success Rate
Description: Technical Success defined as successful delivery and release of BSJ003W into the LAA including successful recapture and retrieval if necessary.
Time Frame: Implant Day
Population: Data collected from Roll-in subjects was analyzed separately from those data collected from ITT cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Implant (ITT) | Roll-in
Number analyzed (Participants) | 42 | 12
Participants | 42 | 12

8. Other Pre Specified Outcome: Warfarin Discontinuation Rate
Description: Warfarin discontinuation rate per protocol. If the TEE shows adequate seal of the LAA with a jet around the device <= 5mm, warfarin therapy should be discontinued.
  Some patients restarted warfarin therapy due to the reasons other than the status of LAA closure.
Time Frame: 45-day, 6-month, 12-month
Population: Data collected from Roll-in subjects was analyzed separately from those data collected from ITT cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Implant (ITT) | Roll-in
Number analyzed (Participants) | 42 | 12
Participants
  At 45-day | 41 | 12
  At 6-month | 40 | 11
  At 12-month: number analyzed (Participants) | 41 | 11
  At 12-month | 39 | 10

ADVERSE EVENTS:
Time Frame: 2 years
Description: Based on the adverse events reported by the investigational site, the sponsor specific coding has been used to summarize adverse events.
Arm/Group | Implant (ITT) | Roll-in
All-Cause Mortality (participants affected / at risk) | 1/42 | 1/12
Serious Adverse Events (participants affected / at risk) | 13/42 | 6/12
Other Adverse Events (participants affected / at risk) | 31/42 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implant (ITT) (N=42) | Roll-in (N=12)
Dyspnea - Heart Failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Renal (Renal and urinary disorders) | 1 (2) | 0 (0)
Device Thrombus Atrial Facing - Post Procedure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0)
Major Bleed Requiring Transfusion (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Stroke (Ischemic) (Nervous system disorders) | 1 (1) | 1 (1)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pericarditis - Unrelated (Non Study) Procedure Or Device (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 0 (0)
Multiple Heart Failure Symptoms (Cardiac disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain - Other (Cardiac disorders) | 1 (1) | 0 (0)
Cranial Bleed - Without Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (General disorders) | 1 (1) | 0 (0)
Head, Eyes, Ears, Norse, Throat (HEENT) (General disorders) | 1 (1) | 0 (0) — The AE name reported by the site was "Chronic otitis media aggravated".
Heart Failure Symptoms - Unspecified (Cardiac disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Led to Death (General disorders) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Systemic Infection (Infections and infestations) | 1 (1) | 0 (0)
Torsades Des Pointes (Cardiac disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 1 (1) | 0 (0)
Vetricular Tachycardia (VT) / Monomorphic VT (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain - Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implant (ITT) (N=42) | Roll-in (N=12)
Head, Eyes, Ears, Nose, Throat (Heent) (General disorders) | 13 (19) | 6 (11) — This AE term includes some symptoms or events reported by the site; ITT (19) includes Common cold (4), Pharyngitis (2), Vertigo (2), Root fracture (2). Roll-in (11) includes Common cold (6). The remaining AEs were reported in one event each.
Gastrointestinal (Gastrointestinal disorders) | 8 (12) | 1 (3)
Integumentary (Skin and subcutaneous tissue disorders) | 6 (10) | 4 (4)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0 (0)
Neurological (Nervous system disorders) | 4 (5) | 0 (0)
Abnormal Laboratory Values (Investigations) | 3 (4) | 2 (3)
Endocrine (Endocrine disorders) | 3 (3) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Fever and/or Virus (Infections and infestations) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.

DOCUMENTS (2):
  • Study Protocol (2016-11-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT03033134/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT03033134/SAP_001.pdf